CLINICAL TRIAL: NCT01803542
Title: Lung Stereotactic Radiation Therapy for Patients With Non-small Cell Lung Cancer and Other Cancers
Brief Title: Stereotactic Radiotherapy (SBRT) of Lung Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 05-0951-C
Record Dates: First submitted 2010-08-10; First posted 2013-03-04 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer; Metastasis From Other Cancers
Keywords: Non-small Cell Lung Cancer; Stereotactic radiation for Lung Cancer; Cone beam CT for Lung Cancer; PET/CT for Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBRT (Experimental): High dose of radiation will be used to treat tumours.
  Interventions: Radiation: Stereotactic Radiation

INTERVENTIONS:
Radiation: Stereotactic Radiation — Participants will receive high doses of radiation treatment to tumours in the lung for 3 to 10 treatment sessions over a total of about 1 to 2 weeks.

SUMMARY:
The purpose of this institutional protocol is to offer SBRT to selected patients in a controlled environment to refine treatment techniques (including dose/fractionation schedules) and standardize follow-up. SBRT has been in clinical use for over a decade in some institutions and the available data suggest that it can be used safely and with good results. This study will see how effective Stereotactic Body Radiation Therapy is for treating tumours in the lung and how often people have side effects. Radiation therapy is usually given once a day, often for a few weeks. In this study, study participants will receive high doses of radiation treatment to tumours in the lung for 3 to 10 treatment sessions over a total of about 1 to 2 weeks.

Several reports indicate that this therapy might shrink tumours and control the cancer for extended periods of time. Although specialists started to treat patients with SBRT over 10 years ago, it is still used in relatively few cancer centres.

DETAILED DESCRIPTION:
SBRT is an adaptation of the principles and experience gained from stereotactic brain RT. SBRT was developed in the early 90s at the Karolinska Institute in Stockholm, Sweden, and is used as an accepted alternative of treatment for patients with early stage lung cancer in many centers in Japan and a number of centers in Germany,USA and elsewhere. It is also now being used for patients who have lung metastases and extra-thoracic disease (primary or metastatic). Many reports indicate excellent local control (80-90% or higher) and minimal toxicity in well selected patients treated with thoracic SBRT.

SBRT has traditionally had the following features:

1. High doses of radiation, usually in a few large fractions (it is "hypofractionated" compared with standard radiotherapy schedules)
2. Multiple radiation beams coming from different directions in the same plane ('co-planar' beams) as well as from different directions and different planes relative to the patient's body ('non-coplanar' beams)
3. Stereotactic beam placement, in that it is guided by a set of coordinates These coordinates are defined in relationship to the precise location of the tumor, determined from medical imaging (e.g. CT, MRI), rather than to a set of external marks (tattoos) or anatomical landmarks (such as bony structures)

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of malignancy, unless the risks of biopsy are unacceptable and the lesion has grown on serial CT scan and/or is PET positive.
* Eligible patients must have staging studies (e.g. chest radiograph, CT scan, MRI/CT Brain/Bone Scan) identifying them as:
* patients with stage I or II, non-metastatic NSCLC (T1, N0, M0; T2, N0, M0; or T3, N0, M0 chest wall primary tumors only)
* patients with a non-lung primary that is controlled and which has metastasized to the lungs alone, in whom potentially curative surgery would otherwise be an option (e.g. colorectal, breast, sarcoma…etc)
* the subset of patients with limited (low) volume metastatic NSCLC or other primary site tumors whom it is felt may derive benefit from highdose SBRT treatment to the primary or metastatic lung tumor. And in whom other sites of metastatic disease are being treated with the desire to achieve long term control. Lesions must meet size criteria in 4.1.2.1
* Patients who have potentially resectable disease should be considered medically inoperable, or else in the judgement of the thoracic surgeon and lung team, surgery is not considered the preferred management option
* Early stage lung cancer: ≤3 parenchymal lung lesions, Metastatic disease to lungs: ≤5 parenchymal lung lesions
* Patients with early stage primary NSCLC should have hilar or mediastinal lymph nodes that are considered N0 on clinico-radiological grounds (i.e. no clinico-radiological evidence of lymph node spread)
* In patients with early stage primary NSCLC and a co-existing malignancy, the co-existing malignancy must have an expected prognosis better than primary lung lesion
* Adequate lung function to tolerate the planned stereotactic radiation
* Previous conventional RT to mediastinum/lung allowed as long as SBRT is not expected to have a high probability of impairing lung function
* Must be ≥ 18 years of age
* Zubrod performance status must be between 0 and 3
* Women of child bearing potential and male participants must use an effective contraceptive method
* Willing and able to give informed consent

Exclusion Criteria:

* Patients with active systemic, pulmonary or pericardial infection
* No concurrent systemic therapy (chemotherapy, immunotherapy or biological therapy), apart from hormone therapy, is allowed
* History of active auto-immune diseases, including systemic lupus erythematous, rheumatoid arthritis, C.R.E.S.T., systemic sclerosis,scleroderma
* Potential candidate for concurrent chemo-radiation therapy
* Patient enrollment on other studies may be permissible. This will depend on patient and study characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Determine local control in patients treated with SBRT. | 10 years
Determine pattern of relapse in patients treated with SBRT. | 10
Determine survival rates in patients treated with SBRT. | 10

SECONDARY OUTCOMES:
To characterize acute and late toxicity | 10 years
Assess the use of PET/CT in aiding target definition and predicting local response | 10 years
Assess the use of Cone Beam CT for precision imaging of the target and avoidance structures at each treatment | 10 years
Assess the use of 4D-computed tomography (CT) planning to determine Internal Treatment Volume (ITV) and Planning Treatment Volume (PTV) | 10 years
Develop organ motion prediction models | 10 years
Monitor major adverse cardiac events | 10 years
Monitor all-cause mortality | 10 years
Monitor cancer specific mortality | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: John Cho, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, University Health Network, Toronto, Ontario, Canada